CLINICAL TRIAL: NCT06901934
Title: JAM3 as a Prognostic Biomarker in Muscle-Invasive Urothelial Carcinoma: Correlation With Therapeutic Response and Survival Outcomes
Brief Title: JAM3 as a Prognostic Biomarker in Muscle-Invasive Urothelial Carcinoma: Correlation With Therapeutic Response, and Survival Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Zeinab Yahia Zaki (Other)
Responsible Party: Sponsor-Investigator, Zeinab Yahia Zaki, zeinab yahia zaki, Assiut University
Organization: Assiut University (Other)
Other Study IDs: JAM3 biomarker bladder cancer
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma Bladder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: junctional adhesion molecule3 expression by immunhistochemistry — * Data record of patient will be reviewed for the following:
  * Clinical features:
  * Age
  * Performance status
  * Risk factors(smoking,stones or bilharziasis)
  * Comorbidities
  * Family history
  * Pathological features:
  * Histological subtype
  * Grade
  * Muscle invasion
  * Carcinoma in situ
  * Immunohistochemistry(IHC):
  JAM3 expression by IHC
  * TNM staging
  * Number of chemotherapy cycles received
  * Radical surgery or
  * CCRT and type of concurrent
  * Post treatment histological response
  * . Follow-Up and Survival Analysis:
  * During treatment: Monitoring for adverse events of chemotherapy and clinical response.
  * After treatment: Imaging and clinical examination every 3 months for 2 years.
  * Correlation of JAM3 expression with progression-free survival (PFS) and overall survival (OS)..

SUMMARY:
Bladder cancer(BC) is the 10th most common cancer globally, with a higher incidence in males than females, being the 6th most common cancer in men with high mortality, causing a societal burden worldwide.

Known risk factors include age, gender, cigarettes, genetic factors, and other environmental influences .

BC can be classified into non-muscle-invasive BC (NMIBC) and muscle-invasive BC (MIBC) . MIBC exhibits a more aggressive nature, correlates with a higher level of T-stage, and has more significant genetic heterogeneity .

Despite comprehensive treatment regimens comprising neoadjuvant chemotherapy, radical cystectomy (RC) and adjuvant immunotherapies, a significant proportion of MIBC patients continue to progress to more advanced stages with limited clinical indicators.

Unfortunately, the mechanisms underlying BC initiation, proliferation, and progression remain largely unknown.

The occurrence of genetic alterations is believed to be closely linked to BC tumorigenesis. Therefore, investigating the genetic alterations might offer opportunities to further understand biological changes in BC .

A key mechanism underlying tumor progression and metastasis is the epithelial-mesenchymal transition (EMT), which is associated with increased invasiveness, chemoresistance, and immune evasion.

EMT is characterized by the downregulation of epithelial markers such as E-cadherin (CDH1) and the upregulation of mesenchymal markers like N-cadherin (CDH2), vimentin, Snail, and ZEB proteins .

Emerging evidence suggests that junctional adhesion molecule 3 (JAM3) plays a role in EMT and cancer progression, with documented involvement in gastric cancer.

However, its significance in MIBC remains poorly understood. Investigating JAM3 expression in MIBC may provide novel prognostic insights and help refine patient stratification for NAC and immunotherapy.

Aim:

This study aims to analyze JAM3 expression in transurethral biopsies from MIUC patients and correlate it with:

* Tumor aggressiveness (grading, staging, and histological features).
* Response to neoadjuvant chemotherapy .
* Patient survival and disease progression.

This study will provide a better understanding of JAM3's role in EMT and MIUC progression, offering potential biomarker-driven insights for treatment stratification.

If JAM3 is validated as a prognostic factor, it could guide personalized therapeutic approaches and optimizing NAC outcomes.

ELIGIBILITY:
Inclusion criteria

1. Patients above 18 years
2. Histopathological confirmed TCC
3. Patients with MIBC
4. Patients eligible for neoadjuvant chemotherapy

Exclusion criteria

1. Patients with metastatic disease
2. Patients ineligible for systemic therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: :Patients diagnosed with muscle invasive urothelial carcinoma( MIUC) and eligible for neoadjuvant chemotherapy( NAC)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The response to neoadjuvant chemotherapy in muscle invasive bladder cancer in relation to JAM3 expression | from enrollment to the end of treatment at 5 months

REFERENCES:
- [Background] Steiner L, Eldh M, Offens A, Veerman RE, Johansson M, Hemdan T, Netterling H, Huge Y, Abdul-Sattar Aljabery F, Alamdari F, Liden O, Sherif A, Gabrielsson S. Protein profile in urinary extracellular vesicles is a marker of malignancy and correlates with muscle invasiveness in urinary bladder cancer. Cancer Lett. 2025 Jan 28;609:217352. doi: 10.1016/j.canlet.2024.217352. Epub 2024 Nov 23. PMID 39586489